CLINICAL TRIAL: NCT01762098
Title: Prevalence of Chronic Endometritis in Patients With Recurrent Miscarriages or Repeated Implantation Failures in In-vitro Fertilization
Brief Title: Chronic Endometritis in Patients With Recurrent Miscarriages or Repeated Implantation Failures in In-vitro Fertilization
Status: Completed | Type: Observational
Sponsor: Clinique Ovo (Industry)
Responsible Party: Sponsor
Other Study IDs: OVO-12-20
Record Dates: First submitted 2013-01-03; First posted 2013-01-07 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Infertility; Endometritis; Abortion, Spontaneous
Keywords: In vitro fertilization; Hysteroscopy; Endometrial biopsy
MeSH Terms: conditions — Infertility; Endometritis; Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Recurrent miscarriages
- Repeated embryo implantation failures

SUMMARY:
Chronic endometritis is a persistent inflammation of the endometrium. Chronic endometritis is asymptomatic or little symptomatic. Sometimes, patient with chronic endometritis can have genital bleeding, pelvic chronic pain, pain during sexual relations, persistent vaginal white loosing. The hysteroscopy can detect the presence or absence of chronic endometritis.

Some studies showed that the endometritis could have an impact on the embryo implantation and could explain recurrent miscarriages or repeated embryo implantation failures.

The goal of this study is to evaluate the frequency of the chronic endometritis in patients with recurrent miscarriages or repeated embryo implantation failures

ELIGIBILITY:
Inclusion Criteria:

Group repeated miscarriages

* Women aged 18 to 43 years
* ≥ 2 miscarriages before 14 weeks of gestation
* Genetic (karyotype x2), thrombophilic and endocrine assessment should be completed

Group of implantation failure in In-vitro fertilization

* Women aged 18 to 45 years
* Absence of pregnancy after 3 good quality embryos transferred in women under 35 years and 4 embryos in the 35 years and over.

Exclusion Criteria:

* Positive pregnancy test
* Unexplained bleeding
* Incomplete miscarriage assessment
* Uterine malformation
* Antibiotic treatment during or within one month prior to the biopsy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Population with recurrent miscarriage or repeated embryo implantation failures.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-11; Primary Completion 2014-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Rate of chronic endometritis | 1 day

SECONDARY OUTCOMES:
Pregnancy rate | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Emmanuel Bouet, MD, Principal Investigator — Université de Montréal
Locations (1):
- Clinique Ovo, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Bouet PE, El Hachem H, Monceau E, Gariepy G, Kadoch IJ, Sylvestre C. Chronic endometritis in women with recurrent pregnancy loss and recurrent implantation failure: prevalence and role of office hysteroscopy and immunohistochemistry in diagnosis. Fertil Steril. 2016 Jan;105(1):106-10. doi: 10.1016/j.fertnstert.2015.09.025. Epub 2015 Oct 9. PMID 26456229